CLINICAL TRIAL: NCT06900686
Title: A Retrospective Study of the Effect of PD-1 Inhibitors in Improving Clinical Outcome for Colorectal Cancer.
Brief Title: Clinical Application of PD-1 Inhibitor in Colorectal Cancer for Improving Survival
Status: Completed | Type: Observational
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: GIHSYSU-RS-01
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2023-03

CONDITIONS: Rectal Cancer; Colon Cancer
Keywords: pd1
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: PD1 Inhibitor — PD1 Inhibitor

SUMMARY:
This trial is a single-center retrospective study. Eligible patients receiving PD-1 inhibitor treatment will enrolled.

DETAILED DESCRIPTION:
In patients with colorectal cancer (CRC), curative surgery combined with chemotherapy ( FOLFOX or CAPOX regimens) has become the standard treatment. However, 20 to 30% of these patients will develop distant metastasis, which ultimately results in death. Oxaliplatin- and fluoropyrimidine-based doublet chemotherapy does not adequately meet the clinical need for tumor shrinkage and downstaging. There is an urgent need to explore drugs with different mechanisms of action in combination with chemotherapy to improve efficacy. Relatively few trials of preoperative therapy have been reported, In recent years, the emergence of immune checkpoint inhibitors has revolutionized cancer treatment. Given the limitations of current treatment strategies in achieving optimal clinical outcomes, this retrospective study aims to research the disease-free survival rates and overall survival (OS) in CRC patients using PD-1 inhibitors.

ELIGIBILITY:
:

Inclusion Criteria:

Willing and able to provide written informed consent. Histological or cytological documentation of adenocarcinoma of the colorectal. Eastern Cooperative Oncology Group's (ECOG) performance status of 0 or 1. CT or MRI scans (done within 30 days of registration) of the chest, abdomen, and pelvis all without clear evidence of distant metastatic (M1) disease.

No clinically significant obstruction, perforation, or bleeding related to the primary tumor.

No previous systemic anticancer therapy for colon cancer disease. Adequate bone marrow, hepatic, and renal function as assessed by the following laboratory requirements conducted within 7 days of starting the study treatment

Exclusion Criteria:

Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years before randomization.

Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.

Heart failure grade III/IV (NYHA classification). Unresolved toxicity higher than CTCAE v.5.0 Grade 1 attributed to any prior therapy/procedure.

Subjects with known allergy to the study drugs or any of its excipients. Current or recent (within 4 weeks before starting study treatment) treatment of another investigational drug or participation in another investigational study.

Breast-feeding or pregnant women Lack of effective contraception.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CRC patients receiving PD-1 inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
DFS | 3years
  disease-free survival

IPD SHARING:
Plan to Share IPD: No